CLINICAL TRIAL: NCT02571907
Title: Clinical Study to Evaluate the Safety and Effectiveness of the Zenith® Branch Endovascular Graft-Iliac Bifurcation
Brief Title: PRESERVE-Zenith® Branch Endovascular Graft-Iliac Bifurcation Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Research Incorporated (Industry)
Responsible Party: Sponsor
Organization: Cook Group Incorporated (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-625 P2
Expanded Access: NCT02475798 (No longer available)
Record Dates: First submitted 2015-09-28; First posted 2015-10-08 (Estimated); Results first posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Aortoiliac Aneurysms; Iliac Aneurysms
Keywords: Zenith aortoiliac aneurysm; Iliac aneurysm; Branch; Connections; Endovascular graft; Graft-iliac bifurcation; Aneurysm; Vascular Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Iliac Aneurysm; Aneurysm; Vascular Diseases; Cardiovascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Zenith® Branch Endovascular Graft-Iliac Bifurcation (Experimental): Zenith® Branch Endovascular Graft-Iliac Bifurcation in combination with the Atrium iCAST™ and the Zenith® Flex AAA Endovascular Graft
  Interventions: Device: Zenith® Branch Endovascular Graft-Iliac Bifurcation,; Device: Atrium iCAST™; Device: Zenith® Flex AAA Endovascular Graft

INTERVENTIONS:
Device: Zenith® Branch Endovascular Graft-Iliac Bifurcation, — Implantation of the Zenith® Branch Endovascular Graft-Iliac Bifurcation.
  Other Names: Branch Graft
Device: Atrium iCAST™ — Implantation of Atrium iCAST
Device: Zenith® Flex AAA Endovascular Graft — Implantation of the Zenith Flex Endovascular Graft

SUMMARY:
The purpose of this extended study is to evaluate the safety and effectiveness of the Zenith® Branch Endovascular Graft-Iliac Bifurcation in combination with the commercially available Atrium iCAST™ covered stent in patients in a treatment of aortoiliac and iliac aneurysms.

ELIGIBILITY:
Inclusion Criteria:

* An aortioiliac or iliac aneurysm
* An unsuitable distal sealing site for a traditional Zenith iliac leg graft within the common lilac artery

Exclusion Criteria:

* Less than 18 years of age
* Inability or refusal to give informed consent
* Disease considerations that would compromise patient safety or study outcomes
* Pregnant, breast-feeding or planning on becoming pregnant prior to completion of the study
* Unwilling or unable to comply with the follow-up schedule
* Simultaneously participating in another investigative device or drug study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2020-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: W. Anthony Lee, MD FACS, Principal Investigator — Christine E. Lynn Heart and Vascular Institute
Locations (28):
- United States (28):
  - Mayo Foundation for Medical Education and Research, Phoenix, Arizona
  - VA Palo Alto HCS, Palo Alto, California
  - Stanford University Medical School, Stanford, California
  - Christine E. Lynn Heart and Vascular Institute, Boca Raton, Florida
  - South Florida Medical Imaging, Fort Lauderdale, Florida
  - University of Florida, Gainesville, Florida
  - Emory University Hospital, Atlanta, Georgia
  - St. Anthony's Medical Center, Rockford, Illinois
  - Methodist Hospital of Indiana, Indianapolis, Indiana
  - University of Kentucky Hospital, Lexington, Kentucky
  - University of Massachusetts, Worcester, Massachusetts
  - William Beaumont Hospital, Royal Oak, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital East Communities, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - UT Southwestern, Dallas, Texas
  - University of Virginia, Charlottesville, Virginia
  - Aurora St. Luke's Hospital, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided
Cook Research Incorporated (CRI) is fully committed to supporting the principles of responsible data sharing, including providing qualified scientific researchers access to deidentified, patient-level data from CRI clinical studies to conduct legitimate scientific research. Data underlying the results reported in this clinical study will be made available for request immediately after approval or clearance of the product and ending 5 years after approval or clearance. Interested researchers may review the "Cook Research Incorporated Policy on Access to Clinical Study Data" at https://www.cookresearchinc.com/extranet/data-access.html and submit a complete research proposal to request data access. Additional study documents (such as the study protocol) will be shared as needed if the data access request is granted. A data sharing agreement will be executed for access to deidentified patient-level data.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zenith® Branch Endovascular Graft-Iliac Bifurcation
Started | 40
Completed | 30
Not Completed | 10
Not completed — Death | 4
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Zenith® Branch Endovascular Graft-Iliac Bifurcation
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American or Black | 3
  Asian | 1
  Hispanic or Latino | 1
  White | 35
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Freedom From Patency-related Intervention Defined as a Secondary Intervention to Treat a > 60 % Stenosis of the Internal Iliac Artery Associated With Clinical Symptoms.
Time Frame: 6 months
Population: One patient died prior to the 6-month visit and thus did not contribute data to the primary outcome. This death was related to a pre-existing condition.
Measure: Count of Participants; unit: Participants
Arm/Group | Zenith® Branch Endovascular Graft-Iliac Bifurcation
Number analyzed (Participants) | 39
Participants | 39
Statistical Analysis 1: Comparison: Zenith® Branch Endovascular Graft-Iliac Bifurcation; Test type: Other; A Bayesian beta-binomial model with a Uniform(0, 1) prior was used to compute a 95% credible interval for the proportion of patients meeting the primary endpoint. The lower bound of this credible interval (2.5th percentile of the posterior distribution) was 91.2%, which was greater than the performance goal of 55%

2. Secondary Outcome: Freedom From Morbidity (i.e., Morbidity Index)
Description: Morbidity index based on a composite endpoint of 31 pre-specified measure elements in seven categories (i.e., cardiovascular, pulmonary, renal, bowel, wound, neurologic, and vascular).
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Zenith® Branch Endovascular Graft-Iliac Bifurcation
Number analyzed (Participants) | 40
Participants | 34
Statistical Analysis 1: Comparison: Zenith® Branch Endovascular Graft-Iliac Bifurcation; Test type: Other; A Bayesian beta-binomial model with a Uniform(0, 1) prior was used to compute a 95% credible interval for the proportion of patients meeting the secondary endpoint. The lower bound of this credible interval (2.5th percentile of the posterior distribution) was 70.8%, which was greater than the performance goal of 46%

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Zenith® Branch Endovascular Graft-Iliac Bifurcation
All-Cause Mortality (participants affected / at risk) | 4/40
Serious Adverse Events (participants affected / at risk) | 26/40
Other Adverse Events (participants affected / at risk) | 15/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zenith® Branch Endovascular Graft-Iliac Bifurcation (N=40)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Stent-graft endoleak (General disorders) | 1 (1)
Vascular stent stenosis (General disorders) | 1 (1)
Vascular stent thrombosis (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 2 (2)
Gastrointestinal infection (Infections and infestations) | 1 (1)
Localised infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 4 (4)
Urinary tract infection (Infections and infestations) | 3 (4)
Vascular graft infection (Infections and infestations) | 1 (1)
Central cord syndrome (Injury, poisoning and procedural complications) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (4)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1)
Vascular procedure complication (Injury, poisoning and procedural complications) | 1 (1)
Ammonia increased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 2 (2)
Oxygen saturation decreased (Investigations) | 1 (1)
Troponin I increased (Investigations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle necrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Intraventricular haemorrhage (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (2)
Neurogenic bladder (Renal and urinary disorders) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 1 (1)
Aneurysm (Vascular disorders) | 1 (1)
Arterial thrombosis (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Intermittent claudication (Vascular disorders) | 1 (1)
Peripheral artery aneurysm (Vascular disorders) | 4 (4)
Peripheral ischaemia (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zenith® Branch Endovascular Graft-Iliac Bifurcation (N=40)
Urinary tract infection (Infections and infestations) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 5 (5)
Testicular pain (Reproductive system and breast disorders) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Aortic aneurysm (Vascular disorders) | 2 (2)
Arterial thrombosis (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-05-09): https://cdn.clinicaltrials.gov/large-docs/07/NCT02571907/Prot_000.pdf